CLINICAL TRIAL: NCT01624337
Title: A Randomized, Double Blind, Placebo-controlled Clinical Trial of Monthly DHA-piperaquine for Malaria Prevention in Cambodia.
Brief Title: Malaria Prevention Cambodia
Acronym: MPC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Medication safety concern
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Collaborators: National Centre for Parasitology, Entomology and Malaria Control, Cambodia (Other); Royal Cambodian Armed Forces (Unknown); United States Army Medical Materiel Development Activity (U.S. Federal Agency)
Responsible Party: Principal Investigator, Philip Smith, Chief, Department of Immunology and Medicine, Armed Forces Research Institute of Medical Sciences, Thailand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WRAIR # 1849; A-17057 (Other: US Army Medical Research and Materiel Command)
Record Dates: First submitted 2012-06-17; First posted 2012-06-20 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; Plasmodium vivax
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Malaria, Vivax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA-piperaquine (Experimental): DHA-piperaquine monthly 2 day treatment course
  Interventions: Drug: DHA-piperaquine
- Placebo (Placebo Comparator): Matching placebo control
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DHA-piperaquine — Drug: Dihydroartemisinin piperaquine
  40/320 mg tablets, 9 tablets total Arms: 2 day treatment course (4.5 tablets per day)
  Other Names: Duocotexcin
  Arms: DHA-piperaquine
Drug: placebo
  Arms: Placebo

SUMMARY:
Trial of monthly DHA-piperaquine for malaria prevention in health volunteers.

DETAILED DESCRIPTION:
This is a two arm, randomized, double-blind, placebo controlled cohort study to determine the protective efficacy of a monthly 2 day treatment course of Dihydroartemisinin-Piperaquine (DP) in adult volunteers in malaria endemic areas of Cambodia.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer 18-65 years of age
2. Able to give informed consent
3. Likely to reside in malaria endemic area for the duration of the study
4. Available for follow-up for anticipated study duration, and agrees to participate for the duration of the study
5. Agrees not to seek outside medical care for febrile illness, except in emergency situations, unless referred by study team
6. Authorized by local commander to participate in the study if on active duty

Exclusion Criteria:

1. Known allergy or other contraindication to DHA, piperaquine treatment, and/or primaquine treatment
2. Significant acute comorbidity requiring urgent medical intervention
3. Positive malaria blood smear.
4. Treatment with an antimalarial drug in the past 30 days.
5. Pregnant or lactating female or a female of childbearing age who does not agree to use a highly effective method of birth control during the study
6. Significantly abnormal EKG including a QTcF interval greater than 450ms at baseline (or 470ms for females) using Fridericia's correction
7. Regular current use of known QTc prolonging medications
8. History of sudden cardiac death in an immediate family member, or personal history of known symptomatic coronary artery disease or arrhythmias
9. Judged by the investigator to be otherwise unsuitable for study participation or non-compliant with study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Protective efficacy | 4 months
  To quantify protective efficacy for the prevention of malaria infection in a setting of mixed multidrug resistant P. falciparum and P. vivax malaria, particularly in non-immune volunteers, in two treatment groups - monthly DHA-piperaquine vs. placebo.
  Protective efficacy will be defined by reduction in the incidence of malaria between treatment and placebo groups.

SECONDARY OUTCOMES:
Cardiac safety of piperaquine as determined by QT interval prolongation | 4-5 months
  To document the effect on the electrocardiogram (EKG), particularly the QTc interval, in patients taking repeated monthly treatment courses of DHA-piperaquine.

CONTACTS AND LOCATIONS:
Overall Officials: DAVID SAUNDERS, MD, MPH, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand; Chanthap Lon, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand
Locations (1):
- Anlong Veng Referral Hospital, Anlong Veaeng, Oddar Meancheay, Cambodia

REFERENCES:
- [Background] Manning J, Vanachayangkul P, Lon C, Spring M, So M, Sea D, Se Y, Somethy S, Phann ST, Chann S, Sriwichai S, Buathong N, Kuntawunginn W, Mitprasat M, Siripokasupkul R, Teja-Isavadharm P, Soh E, Timmermans A, Lanteri C, Kaewkungwal J, Auayporn M, Tang D, Chour CM, Prom S, Haigney M, Cantilena L, Saunders D. Randomized, double-blind, placebo-controlled clinical trial of a two-day regimen of dihydroartemisinin-piperaquine for malaria prevention halted for concern over prolonged corrected QT interval. Antimicrob Agents Chemother. 2014 Oct;58(10):6056-67. doi: 10.1128/AAC.02667-14. Epub 2014 Aug 4. PMID 25092702
- [Derived] Vanachayangkul P, Lon C, Spring M, Sok S, Ta-Aksorn W, Kodchakorn C, Pann ST, Chann S, Ittiverakul M, Sriwichai S, Buathong N, Kuntawunginn W, So M, Youdaline T, Milner E, Wojnarski M, Lanteri C, Manning J, Prom S, Haigney M, Cantilena L, Saunders D. Piperaquine Population Pharmacokinetics and Cardiac Safety in Cambodia. Antimicrob Agents Chemother. 2017 Apr 24;61(5):e02000-16. doi: 10.1128/AAC.02000-16. Print 2017 May. PMID 28193647